CLINICAL TRIAL: NCT02279303
Title: Prescription for Better Breast Health
Brief Title: Rx for Better Breast Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Amelie Ramirez, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HSC20140150H
Record Dates: First submitted 2014-10-15; First posted 2014-10-31 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary Intervention (Experimental): Participants will receive individualized anti-inflammatory dietary prescriptions with six monthly workshops (culinary demonstrations, recipes and meal planning) and behavior change cures reinforced through evidence- and theory-based patient navigation, motivational interviewing, and tailored newsletters personalized to individual readiness for change.
  Interventions: Behavioral: Dietary Intervention
- Dietary Control (Active Comparator): Control participants will receive minimal nutritional information at baseline, monthly American Cancer Society survivorship brochures, and two telephone calls prior to assessment appointments.
  Interventions: Behavioral: Dietary Control

INTERVENTIONS:
Behavioral: Dietary Intervention — Participants will receive individualized anti-inflammatory dietary prescriptions with six monthly workshops (culinary demonstrations, recipes and meal planning) and behavior change cures reinforced through evidence- and theory-based patient navigation, motivational interviewing, and tailored newsletters personalized to individual readiness for change.
  Arms: Dietary Intervention
Behavioral: Dietary Control — Control participants will receive minimal nutritional information at baseline, monthly American Cancer Society survivorship brochures, and two telephone calls prior to assessment appointments.
  Arms: Dietary Control

SUMMARY:
This randomized controlled trial will test the impact of a patient-navigated, anti-inflammatory, culinary-based intervention (reinforced by motivational interviewing [MI] and tailored newsletters) on obese (body mass index [BMI] 30+), early-stage (0-IIIA) breast cancer survivors compared to a control group.

DETAILED DESCRIPTION:
The investigators will recruit English-speaking, early-stage breast cancer survivors (N=200) to a two-arm randomized controlled trial (RCT) involving a 2 (group) by 3 (time) repeated measures design. The intervention will stimulate dietary behavior changes using individualized anti-inflammatory dietary prescriptions with six monthly workshops (culinary demonstrations, recipes and meal planning) and behavior change cures reinforced through evidence- and theory-based patient navigation, motivational interviewing, and tailored newsletters personalized to individual readiness for change. Control participants will receive minimal nutritional information at baseline, monthly American Cancer Society survivorship brochures, and two telephone calls prior to assessment appointments. Groups will be compared at baseline and 6- and 12-month follow-up. Dependent measures will include dietary behavior and levels of cancer-associated biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years or older
* Primary diagnosis of breast cancer
* Fluency in English
* B.M.I. >= 30
* Available for follow-up for 12 months

Exclusion Criteria:

* Clinical evidence of metastatic disease
* Not diagnosed with primary breast cancer
* Lack fluency in English
* B.M.I. < 30

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Achieve USDA-recommended dietary intake based on five major food groups | 12 months
  The USDA has published dietary intake guidelines for 5 major food groups. We will create a composite score ("yes" vs. "no") describing whether ss achieve designated levels of dietary intake for all five food groups. We will compare proportions of study and control women achieving this target at 12-month follow-up controlling for baseline values.
Intervention versus Control group comparison of circulating Adipose Stromal Cells (ASCs) at follow-up | 12 months
  We will compare participant (intervention) versus control levels of circulating Adipose Stromal Cells (ASCs) at 12-month follow-up. Participant levels of ASCs will be significantly lower than controls, controlling for baseline values.
Comparison of Interleukin (IL) pro-inflammatory biomarkers | 12 months
  We will compare participant versus control levels of Interleukins IL3, IL6, IL8 at 12-month follow-up. Participant levels of IL3, IL6, and IL8 will be significantly lower than controls, controlling for baseline values.
Comparison of Interleukin (IL) anti-inflammatory biomarkers | 12 months
  We will compare participant versus control levels of Interleukin IL10 at 12-month follow-up. Participant levels of IL10 will be significantly lower than controls, controlling for baseline values.
Comparison of C-Reactive Protein (CRP) | 12 months
  We will compare participant versus control levels of C-Reactive Protein (CRP) at 12-month follow-up. Participant levels of CRP will be significantly lower than controls, controlling for baseline values.
Comparison of Tumor Necrosis Factor-alpha (TNF-alpha) | 12 months
  We will compare participant versus control levels of Tumor Necrosis Factor-alpha (TNF-alpha) at 12-month follow-up. Participant levels of TNF-alpha will be significantly lower than controls, controlling for baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Amelie Ramirez, DRPH, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States